CLINICAL TRIAL: NCT04351256
Title: Thoracic Radiotherapy Plus Durvalumab in Elderly and/or Frail NSCLC Stage III Patients Unfit for Chemotherapy - Employing Optimized (Hypofractionated) Radiotherapy to Foster Durvalumab Efficacy
Brief Title: Thoracic Radiotherapy Plus Durvalumab in Elderly and/or Frail NSCLC Stage III Patients Unfit for Chemotherapy
Acronym: TRADE-hypo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut für Klinische Krebsforschung IKF GmbH at Krankenhaus Nordwest (Other)
Collaborators: Thoraxklinik-Heidelberg gGmbH (Other); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRADE-hypo; 2019-002192-33 (EudraCT Number); AIO-YMO/TRK-0319 (Other: AIO); ESR-18-13893 (Other Grant/Funding Number: AstraZeneca); 2024-513948-28-00 (EU CTIS Number)
Record Dates: First submitted 2020-02-29; First posted 2020-04-17 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: NSCLC, Stage III
Keywords: Durvalumab; Thoracic Radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Intervention Model Description: Durvalumab treatment and Thoracic Radiotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (HYPO group) (Experimental): * Durvalumab at a fixed dose of 1,500 mg as an IV infusion over 1 hour, on day 1, to be repeated every 4 weeks (Q4W) for a maximum of 12 cycles
  * Thoracic radiation therapy (TRT): hypofractionated thoracic radiotherapy consisting of 20 x 2,75 Gy (55 Gy) within 4 weeks (+9 days)
  Interventions: Drug: Durvalumab Injection [Imfinzi]; Radiation: Thoracic Radiotherapy (TRT) hypofractionated
- Arm B (CON group) (Active Comparator): * Durvalumab at a fixed dose of 1,500 mg as an IV infusion over 1 hour, on day 1, to be repeated every 4 weeks (Q4W) for a maximum of 12 cycles
  * Thoracic radiation therapy (TRT): conventional fractions of 30 x 2 Gy (60 Gy) within 6 weeks (+9 days)
  Interventions: Drug: Durvalumab Injection [Imfinzi]; Radiation: Thoracic Radiotherapy (TRT) conventionally

INTERVENTIONS:
Drug: Durvalumab Injection [Imfinzi] — Durvalumab fixed dose of 1,500 mg
Radiation: Thoracic Radiotherapy (TRT) conventionally — Conventionally fractionated TRT consisting of 30 x 2 Gy (60 Gy) within 6 weeks
  Arms: Arm B (CON group)
Radiation: Thoracic Radiotherapy (TRT) hypofractionated — Hypofractionated TRT consisting of 20 x 2,75 Gy (55 Gy) within 4 weeks
  Arms: Arm A (HYPO group)

SUMMARY:
This is a randomized, open-label, multicenter, phase II trial investigating the combination of thoracic radiotherapy plus Durvalumab in patients with locally advanced, unresectable NSCLC (stage III) that are unfit for chemotherapy (e.g. due to age and/or frailty).

DETAILED DESCRIPTION:
This trial investigates the feasibility and treatment efficacy when combining durvalumab treatment with either conventionally fractionated (CON-group) or hypofractionated thoracic radiotherapy (HYPO-group) in previously untreated NSCLC stage III patients prone to radiotherapy only.

A safety lead-in phase with stop-and-go design will precede full enrollment into the HYPO-group.

Tumor tissue as well as blood and stool samples will be collected for future biomarker analysis.

It is hypothesized that TRT combined with concurrent durvalumab administration in patients with unresectable stage III NSCLC, who are not amenable to sequential radio-/chemotherapy

1. is safe and feasible,
2. will improve treatment efficacy by a synergistic effect of checkpoint inhibition and the photon-induction of immunostimulatory pathways.
3. will have an effect on the immunological characteristics of the tumor, the microenvironment, and the systemic immune response, such as upregulation of PD-L1 or secretion of stimulatory cytokines and recruitment and priming of immunocompetent cells, which might then mediate the "abscopal effect" beyond the irradiated targets.

ELIGIBILITY:
Inclusion Criteria:

1. Fully-informed written consent and locally required authorization (European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years.
3. Histologically documented diagnosis of unresectable stage III NSCLC.
4. Non-feasibility of sequential chemo-/radiotherapy as determined by the site's multi-disciplinary tumor board; if there is no tumor board, then this decision will be made by the investigator in consultation with a radiation oncologist, if the investigator is not a radiation oncologist; or by the investigator in consultation with an oncologist, if the investigator is not an oncologist.
5. Fulfills at least one of the following criteria:

   * Performance status (PS) 2 (ECOG scale)
   * ECOG 1 and CCI ≥ 1
   * Age ≥ 70 years
6. Must have a life expectancy of at least 12 weeks.
7. FEV1 ≥ 40%
8. DLCO or DLCO/VA (Hb-corrected, if available) ≥ 40%
9. FVC or VC ≥ 70%
10. At least one measurable site of disease as defined by RECIST 1.1
11. Adequate bone marrow and renal function including the following:

    * Hemoglobin ≥ 9.0 g/dL;
    * absolute neutrophil count ≥ 1.0 x 103/L;
    * platelets ≥75x 109/L;
    * Calculated creatinine clearance ≥30 mL/min as determined by the Cockcroft-Gault equation
12. Adequate hepatic function (with stenting for any obstruction, if required) including the following:

    * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN);
    * AST (SGOT) / ALT (SGPT) ≤ 2.5x institutional ULN
13. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
14. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.
15. The patient is willing and able to comply with the protocol for the duration of the study, including hospital visits for treatment and scheduled follow-up visits and examinations.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study, or during the follow-up period of an interventional study.
2. Participation in another clinical study with an investigational product within 21 days prior to the first dose of the study treatment.
3. Prior immunotherapy or use of other investigational agents, including prior treatment with an anti-Programmed Death receptor-1 (PD-1),anti-Programmed Death-1 ligand-1 (PD-L1), anti-PD-L2, or anti-cytotoxic T-lymphocyte associated antigen-4 (anti-CTLA-4) antibody, therapeutic cancer vaccines.
4. History or current radiology suggestive of interstitial lung disease.
5. Oxygen-dependent medical condition.
6. Any concurrent chemotherapy, investigational product (IMP), biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (eg, hormone replacement therapy) is acceptable.
7. Prior thoracic radiotherapy within the past 5 years before the first dose of study drug.
8. Major surgery (as defined by the Investigator) within 4 weeks prior to enrollment into the study; patients must have recovered from effects of any major surgery. Note: Local non-major surgery for palliative intent is acceptable.
9. Active or prior documented autoimmune or inflammatory disorders (except inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease]; ( including diverticulitis [with the exception of diverticulosis], celiac disease, systemic lupus erythematosus, Sarcoidosis, or Wegener's syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto's disease) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
10. Active, uncontrolled inflammatory bowel disease [e.g. ulcerative colitis or Crohn's disease]. Patients in stable remission for more than 1 year may be included.
11. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, interstitial lung disease, gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
12. History of another primary malignancy except for:

    * Malignancy treated with curative intent and with no known active disease ≥ 3 years before the first dose of IMP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Toxicity (pneumonitis) | up to 35 months
  Toxicity, defined by the occurence of treatment-related pneumonitis grade ≥ 3
Objective response | up to 35 months
  Objective response evaluated at 12 weeks (3 months) after first durvalumab administration according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
treatment-related AEs and SAEs | up to 35 months
  Occurence of treatment-related AEs and SAEs according to CTCAE V5.0
frequency of abnormal laboratory parameters (hematology panel, chemistry panel, Thyroid-stimulating hormone (TSH)) | up to 35 months
  Frequency of abnormal values of laboratory parameters
Progression Free Survival (PFS) | up to 35 months
  PFS according to RECIST 1.1
Duration of Clinical Benefit | up to 35 months
  Duration of Clinical Benefit (Duration of Complete Response (CR), Partial Response (PR), Stable Disease (SD)) according to RECIST 1.1
Metastasis-Free Survival (MFS) | up to 35 months
  Time from the date of allocation / randomization to the date of first observed metastatic lesion (investigator assessment according to RECIST 1.1) or death from any cause
Overall survival | up to 35 months
  time from the date of treatment allocation to the date of death
Quality of Life (FACT-L) | up to 35 months
  measured by FACT-L questionnaire
objective response rate | up to 35 months
  Descriptive sub-group analyses of efficacy in relation to PD-L1 expression levels (<°1% vs ≥°1%)

OTHER OUTCOMES:
Vulnerability assessment based on the G8-screening questionnaire | up to 35 months
  Vulnerability assessment based on the G8-screening questionnaire and its association to survival and outcome

CONTACTS AND LOCATIONS:
Overall Officials: Farastuk Bozorgmehr, Dr. med., Principal Investigator — Dept. of Thoracic Oncology Thoraxklinik at Heidelberg University
Locations (14):
- Germany (14):
  - Universitätsklinikum Aachen, Aachen
  - DRK Kliniken Berlin-Mitte, Berlin
  - Kliniken der Stadt Köln gGmbH, Lungenklinik Merheim, Cologne
  - Universitätsmedizin Göttingen, Göttingen
  - Onkodok GmbH, Gütersloh
  - Thoraxklinik am Universitätsklinikum Heidelberg, Heidelberg
  - Lungenklinik Hemer, Pneumologie und Thorakale Onkologie, Hemer
  - Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Klinikum Ludwigsburg, Ludwigsburg
  - Universitätsmedizin Mainz, Mainz
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Münster
  - Sana Klinikum Offenbach GmbH, Offenbach
  - Pi.Tri-Studien GmbH, Offenburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bozorgmehr F, Chung I, Christopoulos P, Krisam J, Schneider MA, Bruckner L, Mueller DW, Thomas M, Rieken S. Thoracic radiotherapy plus Durvalumab in elderly and/or frail NSCLC stage III patients unfit for chemotherapy - employing optimized (hypofractionated) radiotherapy to foster durvalumab efficacy: study protocol of the TRADE-hypo trial. BMC Cancer. 2020 Aug 26;20(1):806. doi: 10.1186/s12885-020-07264-8. PMID 32842974